CLINICAL TRIAL: NCT02319291
Title: Outcomes of Total Knee Arthroplasty (TKA) Using the Sigma PS150 Primary Total Knee System
Brief Title: PS150 Total Knee Arthroplasty Outcomes Registry
Status: Completed | Type: Observational
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 13004
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: P.F.C. Sigma PS150 RP Total Knee System
  Interventions: Device: P.F.C. Sigma PS150 RP Total Knee System

INTERVENTIONS:
Device: P.F.C. Sigma PS150 RP Total Knee System — Total Knee Arthroplasty - surgical procedure to replace knee with metal implant

SUMMARY:
This registry is intended to evaluate the clinical outcomes of the DePuy P.F.C. Sigma PS150 RP Total Knee System. 200 participants will be enrolled prospectively or retrospectively and the follow up period will be 5 years. Data collection will include Radiographic Analysis, Knee Society Evaluation and Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* Primary total knee replacement for any indication in accordance with the Instructions For Use accompanying the SIGMA PS150 implant.
* Signed Informed Patient Consent

Exclusion Criteria:

* There are no exclusion criteria for this registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients may be considered for inclusion in the registry if they meet the inclusion criteria below.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Implant Survivorship | 5 years
  Lack of revision with revision meaning no removal or replacement of any TKA component.

SECONDARY OUTCOMES:
Knee Society Score - Knee Score | 1, 3 & 5 years
  Descriptive statistics, including change from baseline (post-op minus pre-op)
Knee Society Score - Function | 1, 3 & 5 years
  Descriptive statistics, including change from baseline (post-op minus pre-op)
Pain sub-question of the Knee Society Score | 1, 3 & 5 years
  Descriptive statistics, including change from baseline (post-op minus pre-op)
Flexion | 1, 3 & 5 years
  Descriptive statistics, including change from baseline (post-op minus pre-op)
Extension | 1, 3 & 5 years
  Descriptive statistics, including change from baseline (post-op minus pre-op)
Radiographic Analysis | 1, 3 & 5 years
  Descriptive statistics
Adverse Events | 1, 3 & 5 years
  Type and frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dekkers, MBBS, Principal Investigator — Greenslopes Private Hospital, Brisbane
Locations (4):
- Australia (2):
  - Greenslopes Private Hospital, Greenslopes
  - Northern Orthopaedics, Sydney
- South Korea (2):
  - Gachon University Gil Medical Center, Incheon
  - Jeju National University Hospital, Jeju City